CLINICAL TRIAL: NCT00971789
Title: A Pilot Study of Sirolimus (Rapamycin, Rapamune[Registered Trademark]) in Subjects With Cowden Syndrome or Other Syndromes Characterized by Germline Mutations in PTEN
Brief Title: Sirolimus to Treat Cowden Syndrome and Other PTEN Hamartomatous Tumor Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080151; 08-C-0151; NCT00722449 (obsolete NCT alias)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Cowden's Disease; Hamartoma Syndrome, Multiple
Keywords: Sirolimus; Cowden Syndrome; PTEN Mutation; Hamartoma Syndrome
MeSH Terms: conditions — Hamartoma Syndrome, Multiple | interventions — Fluorodeoxyglucose F18; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus Patients (Experimental): sirolimus 6 mg by mouth loading dose and 2 mg by mouth daily in a 28 day treatment cycle. Patients who do not have cancer take the drug for a total of two cycles (56 days) unless they develop unacceptable side effects. Those who have cancer may continue sirolimus beyond cycle 2 until their disease worsens or they develop unacceptable side effects.
  Interventions: Radiation: fludeoxyglucose F 18; Drug: sirolimus; Other: Clinical Videography

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Fludeoxyglucose is the radioactive material/compound used as an injection to have a PET scan performed.
  Other Names: FDG-18
Drug: sirolimus — sirolimus 6 mg by mouth loading dose and 2 mg by mouth daily in a 28 day treatment cycle. Patients who do not have cancer take the drug for a total of two cycles (56 days) unless they develop unacceptable side effects. Those who have cancer may continue sirolimus beyond cycle 2 until their disease worsens or they develop unacceptable side effects
  Other Names: Rapamune
Other: Clinical Videography — This examination involves testing of cerebellar function that controls movement, balance, and coordination.

SUMMARY:
Background:

People with phosphatase and tensin homolog deleted on chromosome 10 (PTEN) hamartomatous tumor syndromes (PHTS) have a mutation in one of their genes called PTEN that can lead to benign tumors called hamartomas throughout the body. This puts them at increased risk for breast, thyroid and endometrial cancer.

People with a PTEN mutation have increased activity of proteins such as protein kinase B (AKT) and mammalian target of rapamycin (mTOR), which may be responsible for tumor growth and their increased risk of these cancers.

Experiments show that a drug called sirolimus, which is used to prevent the immune system from rejecting transplanted organs, can inhibit cancer cell growth by blocking the mTOR protein.

Objectives:

To test the ability of sirolimus to decrease the activity of proteins that are regulated by mTOR in both benign and cancerous tumor tissue.

Eligibility:

People 18 years of age and older with Cowden syndrome or other PHTS.

Design:

Sirolimus treatment. Patients take sirolimus once a day in 28-day treatment cycles. Patients who do not have cancer take the drug for a total of two cycles (56 days) unless they develop unacceptable side effects. Those who have cancer may continue sirolimus beyond cycle 2 until their disease worsens or they develop unacceptable side effects.

Evaluations. Patients come to the clinic for a history and physical examination on day 1 of every treatment cycle, then every month for the first two months off therapy, and then at 6 and 12 months. In addition, they have the following procedures:

* Positron emission tomography (PET) scan and neuropsychological testing before starting treatment.
* Clinical photography (photographic documentation of skin lesions) before starting treatment. Patients who do not have cancer have repeat photography at 2 and 8 weeks and then, if the lesions shrink or go away while on therapy, again every month for the first 2 months off sirolimus, then at 6 months and 1 year. Patients who have cancer and continue treatment beyond 8 weeks have repeat photography every 8 weeks while on the study.
* Digital dermoscopy (skin lesion examination using a high resolution camera). This is done at the same intervals as clinical photography.
* Multiple biopsies of the skin and lower intestine, and possibly the tumor in patients with cancer, before starting treatment, at 2 weeks of treatment and at 8 weeks of treatment.
* Blood and urine tests every week while on treatment for the first two cycles, then every 4 weeks for patients who continue treatment beyond two cycles.
* Imaging studies, such as computerized tomography (CT), ultrasound or magnetic resonance imaging (MRI) in patients with cancer before starting treatment and again every two cycles to monitor the tumor size and location.

DETAILED DESCRIPTION:
Background:

* PTEN (phosphatase and tensin homolog deleted on chromosome 10) is a tumor suppressor gene whose function is frequently lost through genetic and epigenetic mechanisms in cancer. Loss of PTEN increases activation of the phosphoinositide 3-kinase (PI3K)/Akt/mTOR pathway, which increases cellular proliferation and survival.
* Germline mutations in PTEN are associated with a number of hamartomatous syndromes, of which Cowden Syndrome (CS) is the prototype. The set of syndromes that are defined by germline PTEN mutations has been labeled PTEN Hamartomatous Tumor Syndromes or PHTS.
* Patients with PHTS suffer increased morbidity and mortality. Benign tumors such as hamartomas occur in virtually every organ, most commonly in the skin and the gastrointestinal tract, which prompts frequent monitoring and resection and causes psychological and physical stressors on patients with this condition.
* Cowden syndrome (CS) patients develop thyroid, breast, and endometrial cancers at an earlier age than the general population, and have an overall increased incidence of these cancers compared to the general population. These patients have increased morbidity from heightened surveillance and diagnostic procedures.
* No medical therapies exist for PHTS patients.
* Because tumors from PHTS patients show increased activation of the PI3K/Akt/mTOR pathway, inhibitors of this pathway might have activity in patients with PHTS.
* Sirolimus (rapamycin) is a specific inhibitor of mTOR that is Food and Drug Administration (FDA)-approved and is preferentially effective in cells with mutant PTEN.
* We hypothesize that sirolimus will have activity in patients with PHTS, as measured by biochemical techniques that will assess mTOR inhibition and clinical tests that will assess the growth and metabolism of benign and malignant tumors.

Objectives:

* The primary endpoint will be inhibition of the mTOR pathway in tissues obtained before and after therapy, as assessed using immunohistochemistry in benign as well as malignant tumors.
* Secondary endpoints will include inhibition of the mTOR pathway in peripheral blood mononuclear cells (PBMCs) as assessed by immunoblotting, changes and duration of change in benign or malignant tumor size as assessed by computed tomography (CT), serial digital photography, digital dermoscopy, changes in tumor metabolism as assessed by positron emission tomography (PET), changes in lymphocyte counts, as well as changes in neuropsychological testing.

Eligibility:

-Adult subjects with documented germline PTEN mutations who meet diagnostic criteria for Cowden Syndrome by international criteria.

Design:

* Subjects will undergo biopsy, imaging, photography, dermoscopy, and neuropsychological testing prior to and after a course of therapy with sirolimus to assess the efficacy of treatment.
* This pilot protocol will test sirolimus at an FDA-approved dose (6 mg by mouth (PO) loading dose/ 2mg PO daily) in a group of twenty patients.
* Treatment will last for 56 days (plus 2 - 3 days to allow flexibility for scheduling of follow-up procedures) for PHTS subjects with benign hamartomatous tumors.
* For PHTS subjects with established malignancy, measurement of disease will be performed every other cycle and treatment will continue until disease progression or unacceptable toxicity.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have documented germline phosphatase and tensin homolog deleted on chromosome 10 (PTEN) mutation performed in a Clinical Laboratory Improvement Amendments (CLIA) approved laboratory.
2. Patients must meet clinical criteria for Cowden Syndrome.
3. Patients must have the capacity to provide informed consent and demonstrate willingness to comply with an oral regimen.
4. Patients must have at least 6 sites amenable to biopsy within the skin and/or gastrointestinal (GI) tract and /or accessible malignant tumor (for patients with malignancy) and agree to the biopsy of these sites prior to and following sirolimus administration.
5. Patients do not need to have malignant tumors, but if they do, they must have relapsed or failed to respond to standard therapy, and the patient's current disease state must be one for which there is no known curative therapy. Patients who are diagnosed with cancer as a consequence of initial positron emission tomography (PET)/computerized tomography (CT) scan will be managed according to the flow diagram illustration.
6. Patients must have not received chemotherapy in the 28 days prior to enrollment.
7. Age greater than or equal to 18 years of age.
8. Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
9. An expected survival of greater than or equal to 3 months.
10. Patients must consent to the use of effective barrier-based contraception during the course of treatment and for three months following discontinuation of treatment.
11. Patients must have normal organ and marrow function as defined below:

    * absolute neutrophil count greater than or equal to 1,500/mL.
    * platelets greater than or equal to 100,000/mL.
    * total bilirubin less than 1.5 times upper limit of institutional normal.
    * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT) less than or equal to 2.5 times upper limit of institutional normal.
    * Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 times upper limit of institutional normal.
    * Creatinine less than 1.5 times upper limit of institutional normal.
12. PHTS subjects with benign hamartomatous disease must have controlled fasting low density lipoprotein (LDL) and triglyceride levels as defined by National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) guidelines. Please see section 3.5 for further details.
13. Patients must have recovered from any acute toxicity related to prior treatments, including surgery. Toxicity should be < grade 1 or returned to baseline.
14. If a patient withdraws consent within two weeks of starting study drug, he/she may request to re-enter study at the principal investigators (PI's) discretion by re-signing consent and being re-registered through the Central Registration Office (CRO) using the initial baseline studies. Sirolimus taken during the period on study (prior to withdrawal of consent) will not be considered as prior sirolimus therapy that otherwise would exclude enrollment.

EXCLUSION CRITERIA:

1. Pregnant or lactating women, due to potentially harmful effects of sirolimus on the embryo or fetus or nursing child.
2. Any concurrent therapy with chemotherapeutic agents or biologic agents or radiation therapy.
3. Patients taking immuno-suppressive agents other than prescribed corticosteroids, which must not exceed the equivalent of 20 mg/d of prednisone.
4. Patients that are on the following cytochrome P450 3A4 (CYP3A4) inhibitors and cannot replace these medications with other equivalent medications for the period of the study: protease inhibitors, cyclosporine, fluconazole, itraconazole, ketoconazole, metoclopramide, felodipine, nifedipine, carbamazepine, Phenobarbital, grapefruit juice, and St. John's Wort.
5. Patients who have received live vaccines in the past 30 days.
6. Patients with human immunodeficiency virus (HIV) seropositivity, due to potential drug interactions between sirolimus and anti-retroviral medications, as well as the unknown effects of single agent sirolimus on the immune system in HIV patients.
7. Patients with interstitial lung disease or pneumonitis.
8. Patients with bleeding diathesis.
9. Patients with prior or active pneumocystis jirovecii (PJP) pneumonia.
10. Patients with prior use of rapamycin, a rapamycin analogue, or other mTOR inhibitor.
11. Patients who do not agree to have multiple repeated biopsies performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Li J, Yen C, Liaw D, Podsypanina K, Bose S, Wang SI, Puc J, Miliaresis C, Rodgers L, McCombie R, Bigner SH, Giovanella BC, Ittmann M, Tycko B, Hibshoosh H, Wigler MH, Parsons R. PTEN, a putative protein tyrosine phosphatase gene mutated in human brain, breast, and prostate cancer. Science. 1997 Mar 28;275(5308):1943-7. doi: 10.1126/science.275.5308.1943. PMID 9072974
- [Background] Zhou XP, Loukola A, Salovaara R, Nystrom-Lahti M, Peltomaki P, de la Chapelle A, Aaltonen LA, Eng C. PTEN mutational spectra, expression levels, and subcellular localization in microsatellite stable and unstable colorectal cancers. Am J Pathol. 2002 Aug;161(2):439-47. doi: 10.1016/S0002-9440(10)64200-9. PMID 12163369
- [Background] Zhou X, Hampel H, Thiele H, Gorlin RJ, Hennekam RC, Parisi M, Winter RM, Eng C. Association of germline mutation in the PTEN tumour suppressor gene and Proteus and Proteus-like syndromes. Lancet. 2001 Jul 21;358(9277):210-1. doi: 10.1016/s0140-6736(01)05412-5. PMID 11476841
- [Derived] Komiya T, Blumenthal GM, DeChowdhury R, Fioravanti S, Ballas MS, Morris J, Hornyak TJ, Wank S, Hewitt SM, Morrow B, Memmott RM, Rajan A, Dennis PA. A Pilot Study of Sirolimus in Subjects with Cowden Syndrome or Other Syndromes Characterized by Germline Mutations in PTEN. Oncologist. 2019 Dec;24(12):1510-e1265. doi: 10.1634/theoncologist.2019-0514. Epub 2019 Jul 26. PMID 31350329
- [Derived] Kalin A, Merideth MA, Regier DS, Blumenthal GM, Dennis PA, Stratton P. Management of reproductive health in Cowden syndrome complicated by endometrial polyps and breast cancer. Obstet Gynecol. 2013 Feb;121(2 Pt 2 Suppl 1):461-464. PMID 23344409
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0151.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus Patients
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus Patients
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.54 (15.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Changes in Benign and Malignant Tumor Tissues as Assessed by Immunohistochemistry.
Description: A biochemical change is defined as a decrease in certain protein levels (e.g. P-AKT (phosphorylated AKT), total S6, P-S6, and P-4E-BP1) important in cell growth. These are measured by collecting tissue samples which stained and protein levels are measured under the microscope. Scoring will be based on distribution and intensity of staining. Distribution will be scored as 0 (0%), 1 (1% to 50%), and 2 (51% to 100%) to indicate the percentage of positive cells of interest in a single core. The intensity of the signal will be scored as 1 (weak), 2 (moderate), and 3 (strong). The distribution score and intensity score will be summed into a total score (TS).
Time Frame: Baseline, day 14, and day 56
Population: No patient underwent biopsy after the study treatment, so no such tissue analysis was done.
Arm/Group | Sirolimus Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events
Time Frame: 47 months
Measure: Number; unit: Participants
Arm/Group | Sirolimus Patients
Number analyzed (Participants) | 18
Participants | 17

ADVERSE EVENTS:
Arm/Group | Sirolimus Patients
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 17/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Patients (N=18)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (12)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (5)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (9)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (5)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (3)
Blood/Bone Marrow - Other (anemia) (Blood and lymphatic system disorders) | 1 (1)
CD4 count (Blood and lymphatic system disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (7)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (bloating) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (4)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2)
Hemoglobin (Metabolism and nutrition disorders) | 7 (9)
Hemorrhage, GI::Colon (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC::Sinus (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 4 (5)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (5)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (4)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (4)
Memory impairment (Nervous system disorders) | 1 (1)
Mood alteration::Depression (Nervous system disorders) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (2)
Pain - Other (R/costal vert. angle; R/flank; shoulder) (General disorders) | 2 (3)
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (3)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 4 (4)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (6)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Rigors/chills (General disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 5 (5)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Vascular - Other (venous insufficiency) (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No